CLINICAL TRIAL: NCT03468348
Title: Duloxetine for Acute Post-mastectomy Pain: Placebo Controlled Dose Ranging Study
Brief Title: Duloxetine for Acute Post-mastectomy Pain
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Diab Fuad Hetta, principle investigator, Assiut University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: SECI-IRB-IORG0006563-437
Record Dates: First submitted 2018-03-11; First posted 2018-03-16 (Actual); Last update posted 2020-06-24 (Actual); Status verified 2020-06

CONDITIONS: Acute Pain
Keywords: duloxetine; mastectomy; postoperative pain
MeSH Terms: conditions — Acute Pain; Pain, Postoperative | interventions — Duloxetine Hydrochloride

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- placebo group (Placebo Comparator)
  Interventions: Drug: Duloxetine
- duloxetine 30 (Active Comparator)
  Interventions: Drug: Duloxetine
- duloxetine 60 (Active Comparator)
  Interventions: Drug: Duloxetine
- duloxetine 90 (Active Comparator)
  Interventions: Drug: Duloxetine

INTERVENTIONS:
Drug: Duloxetine — patients scheduled for mastectomy and axillary evacuation for cancer breast will receive orally, 2 hours before the operation either, placebo capsule, duloxetine 30 mg,duloxetine 60 mg or duloxetine 90 mg capsule.

SUMMARY:
The objective of this study is to evaluate the analgesic effect of oral dulexitine tablet (administered 2 h before surgery) as well as the ideal dose for acute postmastectomy pain.

DETAILED DESCRIPTION:
patients undergoing mastectomy with axillary evacuation will be divided to four groups, Placebo group: received placebo capsule Duloxetine 30: received duloxetine 30 mg capsule Duloxetine 60: received duloxetine 60 mg capsule Duloxetine 90: received duloxetine 90 mg capsule the study medication is administered orall 2 h before surgery. Primary outcome variable: the first postoperative 24 h morphine consumption Secondary outcome: the VAS pain score measured every 4 h in the first 24 h postoperatively.

ELIGIBILITY:
Inclusion Criteria:

* Adult females scheduled for unilateral MRM with axillary evacuation for breast cancer,
* American Society of Anesthesiologists physical status (ASA) class I and II

Exclusion Criteria:

* Patients with a known allergy to Duloxetine or morphine,
* A history of drug or alcohol abuse,
* Patients with impaired kidney or liver functions,
* Patients with chronic pain or regularly receiving analgesics,
* Any psychiatric illness that would interfere with the perception and the assessment of pain.
* Any reason that resulted in the protocol violation.

Ages: 20 Years to 70 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 88 (Actual)
Dates: Start 2018-04-01 (Actual); Primary Completion 2020-02-10 (Actual); Study Completion 2020-02-10 (Actual)

PRIMARY OUTCOMES:
the first postoperative 24 h (patient controlled analgesia [PCA])morphine consumption | the first postoperative 24 hour
  the cumulative patient controlled analgesia morphine consumption required by the patients to relieve their pain in the first postoperative 24 h

SECONDARY OUTCOMES:
The intensity of pain measured by visual analogue pain scale (VAS) | The outcome will be assessed at 0 hour, 2 hour, 4 hour,8 hour, 16 hour and 24 hour postoperatively.
  The intensity of pain measured by visual analogue pain scale (VAS) in which 0 = no pain and 10 = the maximum imaginable pain
The quality of postoperative recovery, assessed by "The QoR-40 questionnaire" (the quality of recovery-40 questionnaire) | the questionnair will be assessed once, 24 hour postoperatively
  It measures five components of patient recovery: physical comfort (12 questions), physical independence (5 questions), emotional state (9 questions), psychological support (7 questions), and pain (7 questions). The sum of each component generates an aggregate score that ranges from 40 (i.e., extremely poor quality of recovery) to 200 (i.e., excellent quality of recovery)
The level of consciousness assessed by "the Modified Ramsay Sedation score" | the score will be measured at 8 hour, 16 hour and 24 hour postoperatively
  awake levels were: I = anxious, agitated, or restless; II = cooperative, oriented, and tranquil; III = responds to command, and asleep levels were dependent on patient's response to a light glabellar tap or loud auditory stimulus; IV= brisk response; V = a sluggish response; and VI = no response)
The occurrence of vomiting | The outcome will be obtained once 24 hour postoperatively
  vomiting is forceful discharge of stomach contents

CONTACTS AND LOCATIONS:
Locations (1):
- Diab, Asyut, Assuit, Egypt

REFERENCES:
- [Derived] Hetta DF, Elgalaly NA, Hetta HF, Fattah Mohammad MA. Preoperative Duloxetine to improve acute pain and quality of recovery in patients undergoing modified radical mastectomy: A dose-ranging randomized controlled trial. J Clin Anesth. 2020 Dec;67:110007. doi: 10.1016/j.jclinane.2020.110007. Epub 2020 Aug 22. PMID 32847776